CLINICAL TRIAL: NCT03163173
Title: A Study to Investigate the Absorption, Metabolism, Excretion, and Mass Balance of GC4419 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galera Therapeutics, Inc. (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GTI-4419-001
Record Dates: First submitted 2017-05-15; First posted 2017-05-22 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers; Healthy
Keywords: Healthy Adult; Superoxide Dismutase; Absorption; Metabolism; Elimination; Mass Balance; Male Subjects
MeSH Terms: interventions — avasopasem manganese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm - Treatment Group (Experimental): 30 mg (~100 μCi) dose of [14C]GC4419 administered as an IV infusion over 15 minutes on Day 1 following an overnight fast
  Interventions: Drug: GC4419

INTERVENTIONS:
Drug: GC4419 — 30 mg (~100 μCi) dose of [14C]GC4419

SUMMARY:
GC4419 is being studied to treat and prevent oral mucositis (painful inflammation) in cancer patients who receive radiation and chemotherapy.

In this study, GC4419 will be mixed with a small amount of radioactive material in order to find out how much study drug is in the blood and to see how the drug is processed and eliminated from the body. The safety and how subjects tolerate the study drug will also be studied.

DETAILED DESCRIPTION:
This is an open-label, single-dose, 1-period study.

On Day 1, a single 30 mg (~100 μCi) dose of [14C]GC4419 will be administered as an IV infusion over 15 minutes. Blood, urine, and fecal samples will be collected to measure total radioactivity (plasma, whole blood, urine, and fecal samples), for GC4419 and its metabolites GC4520 and GC4570 concentrations (plasma, urine, and fecal samples), and for metabolic profiling (plasma, urine, and fecal samples), as total amounts of radioactivity allow, for at least 168 hours postdose (Day 8).

If discharge criteria are not met on Day 8, collection of blood will be collected approximately every 72 hours, and urine and feces collection will continue in 24-hour intervals thereafter (for determination of total radioactivity and metabolic profiling only) until the discharge criteria are met or up to a maximum stay of 28 days (Day 29).

The clinic will attempt to contact all subjects (including subjects who terminate the study early) using their standard procedures approximately 14 days after the last sample collection to determine if any adverse event has occurred since the last sample collection.

Six (6), healthy, adult, non tobacco using, male subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male, 19-55 years of age, inclusive, at screening.
2. Continuous non-smoker who has not used nicotine containing products for at least 3 months prior to dosing and throughout the study.
3. Body mass index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2 at screening.
4. No clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs
5. A non-vasectomized subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond dosing.
6. Must agree not to donate sperm from dosing until 90 days after dosing.
7. Be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated
2. History or presence of clinically significant medical or psychiatric condition or disease
3. History or presence of alcoholism or drug abuse within the past 2 years prior to dosing.
4. History or presence of hypersensitivity or idiosyncratic reaction to the study drug or related compounds.
5. Regularly has less than 1 bowel movement every 2 days.
6. Recent history (within 2 weeks of Day 1) of abnormal bowel habits
7. Positive results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
8. Blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg
9. Heart rate is lower than 40 bpm or higher than 99 bpm
10. Unable to refrain from or anticipates the use of any drug, including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to dosing and throughout the study.
11. Has been on a diet incompatible with the on study diet
12. Donation of blood or significant blood loss within 56 days prior to dosing.
13. Plasma donation within 7 days prior to dosing.
14. Has received radiolabeled substances or has been exposed to radiation sources over the past 12 months or is likely to receive radiation exposure or radioisotopes within the next 12 months such that participation in this study would increase their total exposure beyond the recommended levels considered safe
15. Participation in another clinical study within 28 days prior to dosing.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2017-10-13 (Actual); Study Completion 2017-10-13 (Actual)

PRIMARY OUTCOMES:
Mass balance of GC4419 | From dosing until discharge criteria are met [up to a maximum stay of 28 days postdose (Day 29)]
  Total radioactivity found in biological specimens
Total radioactivity in plasma (AUC0-t) | From dosing until discharge criteria are met [up to a maximum stay of 28 days postdose (Day 29)]
  The area under the concentration time or concentration equivalent time curve, from time 0 to the last observed non-zero concentration (Ct)
Major metabolites in biological specimens. | From dosing until discharge criteria are met [up to a maximum stay of 28 days postdose (Day 29)]
  Total concentrations of GC4419 and its metabolites found in biological specimens
14C radioactivity in whole blood | From dosing until discharge criteria are met [up to a maximum stay of 28 days postdose (Day 29)]
  Change over time in percentage of 14C radioactivity in whole blood
Total radioactivity in plasma (Cmax) | From dosing until discharge criteria are met [up to a maximum stay of 28 days postdose (Day 29)]
  Maximum observed concentration or concentration equivalent
Total radioactivity in plasma (Tmax) | From dosing until discharge criteria are met [up to a maximum stay of 28 days postdose (Day 29)]
  Time to reach Cmax

CONTACTS AND LOCATIONS:
Overall Officials: Jon T Holmlund, MD, Study Chair — Galera Therapeutics
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No